CLINICAL TRIAL: NCT05331183
Title: A Phase 3 Open-label Study Evaluating the Long-term Safety and Efficacy of Elexacaftor/Tezacaftor/Ivacaftor in Cystic Fibrosis Subjects With Non-F508del CFTR Genotypes
Brief Title: Study to Evaluate Elexacaftor/Tezacaftor/Ivacaftor (ELX/TEZ/IVA) Long-term Safety and Efficacy in Subjects Without F508del
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX21-445-125; 2021-005914-33 (EudraCT Number); 2024-515637-14-00 (Other: EU Trial (CTIS) Number)
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — elexacaftor, ivacaftor, tezacaftor drug combination; ivacaftor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ELX/TEZ/IVA (Experimental): Part A: Participants will receive ELX/TEZ/IVA in the morning and IVA in the evening for 96 weeks.
  Part B: Participants will receive ELX/TEZ/IVA in the morning and IVA in the evening for an additional 96 weeks.
  Interventions: Drug: ELX/TEZ/IVA; Drug: IVA

INTERVENTIONS:
Drug: ELX/TEZ/IVA — Fixed-dose combination (FDC) tablets for oral administration.
  Other Names: VX-445/VX-661/VX-770; elexacaftor/tezacaftor/ivacaftor
Drug: IVA — Tablets for oral administration.
  Other Names: VX-770; ivacaftor

SUMMARY:
This study will evaluate the long-term safety, efficacy and pharmacodynamics of ELX/TEZ/IVA in participants with cystic fibrosis (CF) with at least 1 non-F508del ELX/TEZ/IVA-responsive CF transmembrane conductance regulator (CFTR) gene mutation.

ELIGIBILITY:
Key Inclusion Criteria:

Part A: Completed study drug treatment in parent study or had study drug interruption(s) in parent study but completed study visits up to the last scheduled visit of the treatment period in the parent study

Part B: Completed study drug treatment in Part A or had study drug interruption(s) in Part A but completed study visits up to the last scheduled visit of the treatment period of Part A

Key Exclusion Criteria:

History of study drug intolerance in the parent study

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2022-11-23 (Actual); Primary Completion 2027-04-06 (Estimated); Study Completion 2027-04-06 (Estimated)

PRIMARY OUTCOMES:
Parts A and B: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 up to Week 196

SECONDARY OUTCOMES:
Part A: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 second (ppFEV1) | From Baseline up to Week 96
Part A: Absolute Change in Sweat Chloride (SwCl) | From Baseline up to Week 96
Part A: Absolute Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain (RD) Score | From Baseline up to Week 96
Part A: Absolute Change in Body Mass Index (BMI) | From Baseline up to Week 96
Part A: Absolute Change in Weight | From Baseline up to Week 96
Part A: Number of Pulmonary Exacerbations (PEx) | From Baseline up to Week 96

CONTACTS AND LOCATIONS:
Locations (81):
- Medizinische Universität Innsbruck - Heilstättenschule Universitätsklinik, Innsbruck, Austria
- Belgium (6):
  - CUB Hôpital Erasme, Brussels
  - UZ Brussel - Campus Jette, Brussels
  - Universitair Ziekenhuis Antwerpen (UZA) - Antwerp University Hospital, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
  - Universite Catholique de Louvain - Pulmonology, Woluwe-Saint-Lambert
- Canada (6):
  - Stollery Children's Hospital, Edmonton
  - Le Centre de recherche du CHUM (CRCHUM), Montreal
  - McGill University Health Centre, Glen Site, Montreal Children's Hospital, Montreal
  - Hospital for Sick Children - Pulmonology, Toronto
  - British Columbia Children's Hospital, Vancouver
  - St. Paul's Hospital - Pulmonology, Vancouver
- Czechia (2):
  - Klinika Detskych Infekcnich Nemoci, Brno
  - Motol University Hospital, Prague
- France (16):
  - Hopital Femme Mere-Enfant, Bron
  - Centre Hospitalier Intercommunal Creteil - Pulmonology, Créteil
  - Institut Cœur Poumon, CHU de Lille, Lille
  - Hopital Nord, Marseille
  - Hopital Arnaud de Villeneuve - Service de Pneumologie et Maladies Respiratoires, Montpellier
  - Hôpital Nord Laennec, Nantes
  - CHU de Nice - Hôpital Pasteur 2, Nice
  - Hopital Cochin - Pulmonology, Paris
  - Hopital Necker Enfants Malades - Pulmonology, Paris
  - Hopital Robert Debre - Pulmonology, Paris
  - Hôpital Lyon Sud - Pulmonology, Pierre-Bénite
  - Hôpital américain de Reims - Département de pédiatrie A, Reims
  - Hôpital Sud - Rennes, Rennes
  - Centre de Perharidy, Roscoff, Roscoff
  - Hopital Larrey, Toulouse
  - Hopital Bretonneau, Tours
- Germany (14):
  - Charité - Paediatric Pulmonology Department, Berlin
  - University Hospital Cologne (Koeln) - CF-Studienzentrum, Cologne
  - Ruhrlandklinik, Essen
  - Klinikum der Johann-Wolfgang-Goethe Universitaet - Pulmonology, Frankfurt
  - Justus-Liebig-Universität Gießen, Giessen
  - Universitätsklinikum Halle (Saale) / Universitätsklinik und Poliklinik für Innere Medizin, Schwerpunkt Pneumologie, Halle
  - Medizinische Hochschule Hannover - Clinic for Pediatric Pneumology, Allergology and Neonatology, CF-Centre, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Mukoviszidose-Zentrum am Universitätsklinikum Jena, Jena
  - Johannes Gutenberg-Universitaet, Mainz
  - Dr. von Haunersches Kinderspital - Pulmonology, München
  - Lungenheilkunde Munchen - Pasing, München
  - Klinik für Kinder- und Jugendmedizin, Münster
  - Klinikum Westbrandenburg (CF), Potsdam
- National Koranyi Institute for TBC and Pulmonology, Budapest, Hungary
- Italy (11):
  - Azienda Ospedaliero Universitaria delle Marche, Ancona
  - Azienda Ospedaliero Universitaria Ospedale Meyer, Florence
  - IRCCS Istituto Giannina Gaslini-Ospedale Pediatrico, Genova
  - Policlinico Universitario G. Martino, Messina
  - Fondazione IRCCS Ospedale Maggiore Policlinico, Mangiagalli e Regina Elena, Milan
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliero Universitaria Federico II Napoli, Naples
  - Azienda Ospedaliero Universitaria (AOU) San Luigi Gonzaga, Orbassano
  - Azienda Ospedaliera Regionale 'San Carlo', Potenza, Potenza
  - IRCSS Ospedale Pediatrico Bambino Gesu - Pulmonology, Rome
  - Azienda Ospedaliera di Verona - Ospedale Civile Maggiore, Verona
- Netherlands (5):
  - Amsterdam UMC - locatie AMC - Afdeling Longgeneeskunde, Amsterdam
  - Radboud University Medical Center - Pulmonology, Nijmegen
  - Erasmus Medisch Centrum - Pulmonology, Rotterdam
  - HagaZiekenhuis, The Hague
  - UMCU, Locatie Wilhelmina Kinderziekenhuis, Utrecht
- Oslo University Hospital, Department of Paediatric Medicine, Oslo, Norway
- Poland (2):
  - Pediatric Hospital Polanki named of Maciej Płażyński, Gdansk
  - Instytut Matki i Dziecka, Klinika Mukowiscydozy IMiD, Oddział Chorób Płuc SZPZOZ im.Dzieci Warszawy w Dziekanowie Leśnym, Łomianki
- Unidade Local de Saúde de Santa Maria, E.P.E. - Pulmonology, Lisbon, Portugal
- Spain (12):
  - Hospital de Cruces, Barakaldo
  - Hospital Saint Joan de Deu, Barcelona
  - Hospital Universitari Vall d´Hebron Servicio de Broncoscopia, Barcelona
  - Hospital Universitario de Jerez de la Frontera, Jerez de la Frontera
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - Hospital Universitario 12 de Octubre - Pulmonology, Madrid
  - Hospital Universitario Ramon y Cajal - Pulmonology, Madrid
  - La Paz Infantil, Madrid
  - Hospital Virgen de la Arrixaca, Murcia
  - Institut d´Investigacio i Innovacio Parc Tauli, Sabadell
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario y Politecnico La Fe - Pulmonology, Valencia
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset - Göteborg CF-center, Gothenburg
  - Karolinska University Hospital - Pulmonology, Stockholm
- Kinderspital Zuerich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/our-science/clinical-trials-data-sharing/